CLINICAL TRIAL: NCT02511873
Title: Randomized Crossover Trial of Fycompa in the Treatment of Pain Associated With Small Fiber Neuropathy (SFN)
Brief Title: Fycompa in Subjects With Small Fiber Neuropathy (SFN)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PNA Center for Neurological Research (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Todd Levine, MD, Primary Investigator, PNA Center for Neurological Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FYCOMPA
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Neuropathy, Small Fiber
Keywords: Fycompa; Small Fiber Neuropathy; SFN; Neuropathy; Pain
MeSH Terms: conditions — Small Fiber Neuropathy; Pain | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fycompa (Experimental): Fycompa dose is chosen based on tolerability and efficacy. 2mg to 8mg daily for 6 weeks then washed out.
  Interventions: Drug: Fycompa
- Placebo (Placebo Comparator): Inactive ingredient equal to 2mg tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fycompa — Subjects will take Fycompa for 6 weeks with a dose range of 2mg to 8mg daily
  Other Names: Perampanel; E2007; AMPA - type Glutamate Receptor Antagonist
  Arms: Fycompa
Drug: Placebo — Placebo (looks like study drug but has no active ingredients) for 6 weeks with a dose range of 2mg to 8mg daily
  Arms: Placebo

SUMMARY:
This is a Phase II, 2 arm randomized crossover study. Subjects will be assigned to either active agent or placebo and then crossover to the other arm. This study is designed to evaluate whether Fycompa improves the quality of life in patients with small fiber neuropathy.

DETAILED DESCRIPTION:
This study will enroll 30 patients from our center alone with a proven SFN diagnosis by a skin biopsy assessment of intraepidermal nerve fiber density. The patients must also have a pain score of a least 5 on a VAS Scale. Patients will receive Fycompa 2mg tablets. Each week patients will be allowed to titrate up by 2mgs up to a maximum dose of 8mg a day. This dosing has been used in numerous pain studies when no single dose has been proven to be effective. This does not seem to reduce the validity of the placebo phase. Patients can choose the dose they feel is best tolerated and most efficacious. Once patients choose this dose they will be randomized into two arms. Each arm will last 6 weeks. Such that patient will receive the dose they chose as most efficacious for 6 weeks or matching placebo for 6 weeks. Then each patient will crossover to the other arm. Investigator will assess compliance by counting pills at each visit. This will provide the ability to see which dose most patients prefer and then study the dose in a blinded randomized fashion. There will be 5 office visits and 3 phone visits in the study and . Patients will keep a diary of weekly VAS pain scores.

ELIGIBILITY:
Inclusion Criteria:

1. Small Fiber Neuropathy(SFN) proven by skin biopsy assessment of intraepidermal nerve fiber density.
2. Pain scores of at least a 5 on a VAS scale.
3. Male or Female 18 to 60 years old.
4. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
5. Stable dose of current pain medication or any medication used for SFN 60 days prior to screening.
6. Women of reproductive age must agree to use double-barrier method of contraception.

Exclusion Criteria:

1. History of intolerance or hypersensitivity to Fycompa.
2. History of psychosis, drug or alcohol abuse within the last 2 years.
3. Malignancy within the last 2 years (except skin cancer).
4. Clinically significant condition (including but not limited to cardiovascular or hepatic diseases and seizure disorders).
5. Pregnant females, breastfeeding females, females of childbearing potential not using effective contraception.
6. Subjects with other severe pain conditions which may impair the self-assessment of pain due to SFN.
7. Exclusion medications for this study: Carbamazepine, Carbatrol, Tegretol, Tegretol XR, Equetro, Epitol, Phenytoin, Dilantin, Phenytek, Oxcarbazepine, Trileptal, Rifampin, Refadin, Rimactane and St. John Wort.
8. Subjects with renal impairment or on hemodialysis or who have hepatic impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To Assess the Change of Pain Symptoms Upon Treatment of Fycompa in Comparison to Placebo using Visual Analog Scale (VAS) andBrief Pain inventory(BPI) Short Form | Baseline, Week 5, Week 12 and Week 18

SECONDARY OUTCOMES:
To Assess improvement of Quality of Life Upon Treatment of Fycompa in Comparison to Placebo using Neuro QOL Lower Extremity Function Scale, Patient Global impression of Change (PGIC) Scale and Treatment Satisfaction Questionnaire for Medication (TSQM) | Baseline, Week 5, Week 12 and Week 18

CONTACTS AND LOCATIONS:
Overall Officials: Todd Levine, MD, Principal Investigator — PNA Center for Neurological Research
Locations (1):
- PNA Center for Neurological Research, Phoenix, Arizona, United States